CLINICAL TRIAL: NCT05851092
Title: A Single Arm, Open, Multicenter Phase I Clinical Study on the Safety, Tolerance, and Pharmacokinetics of HRS-2189 Single Drug in Patients With Advanced Malignant Solid Tumors
Brief Title: Phase I Clinical Study of HRS-2189 in the Treatment of Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-2189-I-101
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-04

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-2189 Tablets (Experimental)
  Interventions: Drug: HRS-2189 Tablets

INTERVENTIONS:
Drug: HRS-2189 Tablets — HRS-2189 Tablets

SUMMARY:
This study is a multi center, open label, dose increasing/dose expanding/efficacy expanding phase I clinical trial aimed at evaluating the safety, tolerance, PK characteristics, and anti-tumor efficacy characteristics of HRS-2189 single drug in patients with advanced malignant solid tumors. This study was divided into three stages: dose escalation, dose expansion, and efficacy expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study, sign an informed consent form, have good compliance, and can cooperate with follow-up
2. Age ≥ 18 years old (including boundary value, calculated based on the date of signing informed consent), Male or female
3. ECOG score: 0-1
4. Expected survival ≥ 12 weeks
5. Local recurrent or metastatic advanced malignant solid tumor confirmed by histopathology or cytopathology and not resectable, and currently fails to undergo standard treatment or has no standard treatment plan
6. If enrolled in ER positive and HER2 negative female breast cancer subjects, they need to meet the criteria defined in the guidelines of the American Association of Clinical Oncology/American College of Pathologists
7. Baseline presence of at least one extracranial measurable lesion that meets the RECIST v1.1 standard
8. The functional level of important organs is basically normal, meeting the requirements of the scheme
9. Previous treatment: Before the first medication in this study, the interval between receiving nitrosourea or mitomycin C ≥ 6 weeks; Receiving cytotoxic drugs, endocrine therapy, immunotherapy, targeted therapy, surgical interval (except puncture biopsy or PICC catheterization or PORT infusion port catheterization) or other clinical studies with the last medication ≥ 4 weeks; Interval from the end of radiotherapy ≥ 2 weeks
10. Adverse events caused by other treatments for the subject returned to a severity level of NCI-CTCAE V5.0 ≤ 1 (excluding hair loss and other adverse events judged tolerable by the investigator)
11. Female subjects with fertility must agree to use highly effective contraception during the study treatment period and within 7 months after the last medication; Male subjects must agree to use highly effective contraception during the study treatment period and 4 months after the last medication; Female subjects with fertility must have a negative serum HCG test within 7 days before the first medication in the study, and must be in non lactation. If the serum HCG is weakly positive, it is necessary for the researcher to evaluate and judge it as a non pregnant state, and urine HCG should be tested before medication, with a negative result
12. Volunteer to participate in this clinical trial, willing and able to follow the procedures related to clinical visits and research, understand the research procedures, and have signed informed consent

Exclusion Criteria:

1. Subjects with cancerous meningitis or untreated central nervous system metastasis
2. Uncontrolled pleural, abdominal, and pericardial effusion
3. Clinical symptoms or diseases of the heart that are not well controlled
4. Arterial/venous thrombotic events occurred within 6 months before the first medication administration
5. Active infection or unexplained fever>38.5 ° C occurred within 4 weeks before or on the day of the first medication (subjects with tumor fever are judged by the investigator to be included in the study)
6. Subjects with congenital or acquired immune dysfunction (such as HIV infected persons); Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
7. Subject has active hepatitis
8. Subjects had other malignant tumors within the past 3 years, except for fully treated basal or squamous cell skin cancer or cervical carcinoma in situ
9. Those who are unable to swallow tablets normally or have gastrointestinal dysfunction that may affect drug absorption according to the judgment of the researcher
10. Patients participating in the QT/QTc study have used any medication that has the risk of prolonging the QT/QTc interval or causing torsade de pointe (TdP) within 4 weeks before the first medication, have a previous history of congenital QT interval prolongation syndrome or a family history of QT interval prolongation, have an implanted pacemaker or automatic implantable cardioverter defibrillator, and cannot correct electrolyte disturbances that affect the QT/QTc study
11. Pregnant and lactating women, or planning to become pregnant during the study period
12. According to the judgment of the researcher, the subject has other factors that may lead to the forced termination of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs+SAEs | from the first drug administration to within 30 days for the last treatment dose
Dose limited toxicity (DLT) of HRS-2189 | up to 35 days
Maximum tolerated dose（MTD）of HRS-2189 | up to 35 days
Recommended Phase II Dose (RP2D) of HRS-2189 | up to 35 days

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of HRS-2189: Cmax | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: Tmax | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: AUC0-t | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: AUC0-inf | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: Cmax,ss | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: Tmax,ss | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: Cmin,ss | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: AUCss | 2 months
Evaluation of pharmacokinetic parameter of HRS-2189: Rac | 2 months
Bioavailability of HRS-2189 on an empty stomach and after meals | up to 9 days
Objective Response Rate (ORR) | every 8 weeks since Day 8 administration,an average of 1 year
  Number of responders Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed by CT or MRI
Duration of response (DoR) | every 8 weeks since Day 8 administration,an average of 1 year
  Time from documentation of tumor response to disease progression assessed among patients who had an objective response
Disease control rate (DCR) | every 8 weeks since Day 8 administration,an average of 1 year
  Complete response + Partial response + Stable disease (CR+PR+SD) based on RECIST 1.1
Progression free survival（PFS） | every 8 weeks since Day 8 administration,an average of 1 year
  The time from enrollment to the progression of tumors (in any aspect) or death (for any reason)

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided